CLINICAL TRIAL: NCT04710979
Title: Feasibility of a Yoga Intervention in Sedentary African-American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00010979; R34AT011036 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2021-01-15 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Sedentary Behavior
Keywords: Yoga; African-American; Feasibility Study
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Intervention Group (Experimental)
  Interventions: Behavioral: Yoga Intervention
- Control Group (No Intervention): Control participants will receive no guidance from the research staff to change their behavior.

INTERVENTIONS:
Behavioral: Yoga Intervention — This group will have in-person, 60 minute yoga sessions three times per week for 12 weeks. These sessions will also include a sharing circle to provide group feedback as to how the practice felt and integration into ones' daily life. There will be biweekly themes established for these sessions (i.e. common yoga poses, importance of breath) and biweekly in-person workshops will be offered. These will be specialty classes for participants to experience additional exposure to meditation and breathing. They will be a longer format so participants can delve deeper into yogic philosophy and practice. There will also be a private Facebook group for participants to connect with each other and for the research staff to maintain contact and share information with the participants (eg. weekly reminder for yoga sessions and workshops).
  Arms: Yoga Intervention Group

SUMMARY:
This study aims to test the feasibility, acceptability, safety of a 3-month hatha and restorative yoga intervention to decrease sedentary behavior, stress and blood pressure in sedentary African-American women.

DETAILED DESCRIPTION:
This study aims to assess feasibility of a hatha and restorative yoga intervention compared to a control group. Investigators will examine feasibility of participant recruitment, retention and adherence; fidelity of intervention delivery; and intervention materials. Investigators also aim to evaluate the acceptability and safety of a hatha and restorative yoga intervention compared to a control group. Investigators will examine the acceptability of intervention location and strategies, class format, enjoyment of sessions, and safety of the intervention. Finally, investigators aim to test feasibility and appropriateness of the targeted outcomes for subsequent trials. Expected outcomes will be properly measured, but no comparisons between intervention and control groups will be made.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as an African-American woman at least 18 years old
* Engaging in less than 30 minutes/week of moderate-to-vigorous physical activity
* If employed, working in a sedentary occupation that requires primarily seated work; • If unemployed, typical day involves sedentary, primarily seated activities
* Able to exercise for 20 minutes continuously
* No pre-existing condition that limits physical activity
* Access to a computer (or mobile device) and internet service

Exclusion Criteria:

* Diagnosed with heart disease, diabetes, cancer, kidney, liver disease, major depression or bipolar disease
* Take more than two daily medications for lipids or blood pressure
* Current smoker

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daheia J Barr-Anderson, PhD, MSPH, Principal Investigator — University of Minnesota; Mark A Pereira, PhD, MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the greater Twin Cities, MN area via social media, emails to organizations, flyers, websites, and a news segment on a local TV station. The online interest/pre-screening survey received 319 unique responses between March 2022 and May 2022. The first participant consented and enrolled on May 2, 2022.
Pre-assignment Details: Of the 131 individuals who were assessed for eligibility after pre-screening, 69 met the inclusion criteria and consented. Prior to randomization, 1 participant voluntarily withdrew from the study due to discomfort providing salivary samples. Of the 68 participants randomized to intervention groups, 1 participant involuntarily withdrew prior to the start of the intervention due to injuries sustained in an accident unrelated to the study.
Period: Overall Study
Arm/Group | Yoga Intervention Group | Control Group
Started | 34 (Thirty-four participants were randomized to the yoga intervention group. However, one participant involuntarily withdrew from the study after randomization but prior to the start of the intervention due to injuries sustained in an accident unrelated to the study. Thus, only 33 intervention participants actually started the intervention.) | 34
Post-Intervention | 31 | 26
3-Month Follow-Up | 23 | 28
Completed | 31 | 30
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Intervention Group | Control Group | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (9.4) | 43.4 (11.2) | 44.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 34 | 34 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 34 | 68
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 34 | 68
Education [Count of Participants; unit: Participants] — Highest level of education completed.
  Participants
    Completed high school or GED | 2 | 0 | 2
    Some college or technical school | 6 | 8 | 14
    Completed associate's degree or technical school | 3 | 4 | 7
    Completed bachelor's degree | 8 | 7 | 15
    Attends or has attended graduate school | 3 | 3 | 6
    Completed graduate school | 12 | 12 | 24
Employment [Count of Participants; unit: Participants] — Current occupation status.
  Participants
    Employed | 30 | 31 | 61
    Not currently employed | 2 | 1 | 3
    Student | 2 | 2 | 4
Income [Count of Participants; unit: Participants] — Total household income before taxes in the past year.
  Participants
    <$35,000 | 3 | 5 | 8
    $35,000 - $49,999 | 5 | 6 | 11
    $50,000 - $74,999 | 12 | 9 | 21
    $75,000 - $99,999 | 2 | 4 | 6
    >$100,000 | 10 | 9 | 19
    Prefer not to answer | 2 | 1 | 3
Marital Status [Count of Participants; unit: Participants]
  Married | 13 | 8 | 21
  Not married, living with partner | 3 | 3 | 6
  Separated/Divorced/Widowed | 8 | 7 | 15
  Single, never married | 10 | 16 | 26
Sedentary Behavior [Mean (Standard Deviation); unit: Hours per day] — Average total number of hours per day engaged in sedentary behavior, assessed via participants wearing the activPAL4 micro accelerometer for 7 consecutive days. Population: Activity monitor data missing from four participants who did not return their activity monitors.
  Hours per day
    number analyzed (Participants) | 32 | 32 | 64
    (all) | 10.7 (1.7) | 10.2 (2.0) | 10.5 (1.8)
Systolic and Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Average of three blood pressure readings measured using the OMRON Hem 907XL blood pressure monitor. Population: Unable to obtain blood pressure readings from one intervention participant due to equipment malfunction.
  mmHg
    SBP: number analyzed (Participants) | 33 | 34 | 67
    SBP | 114.2 (13.6) | 116.1 (14.0) | 115.2 (13.8)
    DBP: number analyzed (Participants) | 33 | 34 | 67
    DBP | 77.2 (11.5) | 77.2 (12.7) | 77.2 (12.1)
Perceived Stress [Mean (Standard Deviation); unit: units on a scale] — Measured using the 14-item Perceived Stress Scale. Each item is scored from 1-5, with higher scores indicating higher perceived stress. Estimates represent the mean total score of the 14 items, ranging from 1-5. Scale was included in an online survey that participants completed at the data collection site via an iPad. Survey items asked participants how often they had experienced acute stress within last month.
  units on a scale | 2.9 (0.4) | 2.8 (0.5) | 2.8 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recruited (Feasibility)
Description: Goals were for 200 women recruited and screened for eligibility, and 60 enrolled and consented.
Time Frame: Baseline
Population: Total number of participants who were recruited and screened via an online interest/pre-screening survey. For this outcome measure analysis, we will report the number of recruited participants who then enrolled and consented in the study. This pre-assignment sample size differs from the number of participants who started the 12-week intervention period because 2 participants withdrew from the study before the 12-week intervention period began.
Measure: Count of Participants; unit: Participants
Groups:
- Total Recruitment Sample, Pre-Assignment: All participants who filled out the online pre-screening interest survey, including those were later 1) excluded from the study before assignment to groups due to not meeting eligibility criteria or completing the consent process, and 2) randomly assigned into the yoga intervention group and control group arms.
Arm/Group | Total Recruitment Sample, Pre-Assignment
Number analyzed (Participants) | 319
Participants
  Number of Participants Recruited and Screened | 319
  Number of Participants Enrolled and Consented | 69

2. Primary Outcome: Rate of Participant Retention and Adherence (Feasibility)
Description: At least 80% of intervention participants attend at least 80% of intervention sessions
Time Frame: During the 12-week yoga intervention
Population: The number of participants analyzed was 33 because this outcome was measured during the 12-week yoga intervention and prior to the post-intervention data collection milestone. There were originally 34 participants randomized to the yoga intervention, but 1 intervention participant officially withdrew from the study prior to the start of the intervention. Thus, we calculated attendance rates for 33 intervention participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group
Number analyzed (Participants) | 33
Participants | 8

3. Primary Outcome: Fidelity of Intervention Delivery (Feasibility)
Description: At least 90% (8 of 9 class segments) of each of the 6 videotaped sessions is delivered as planned based on training.
Time Frame: During the 12-week yoga intervention
Population: Please note that no participants were analyzed for this outcome measure. Six video recordings of yoga intervention sessions were analyzed to enumerate the number of yoga segments (e.g., planned specific yoga components) that were completed as a percentage of the total (n = 9 yoga segments per session).
Measure: Count of Units; unit: yoga segments
Units Other Than Participants: yoga segments
Groups:
- Yoga Segments: Six 60-minute yoga sessions were randomly selected from the 72 total yoga intervention sessions to be recorded and analyzed for fidelity. Instructors were trained and expected to teach 9 yoga segments (e.g., planned specific yoga components) within each session.
Arm/Group | Yoga Segments
Number analyzed (Participants) | NA
Number analyzed (yoga segments) | 9
yoga segments
  Session 1 | 8
  Session 2 | 7
  Session 3 | 9
  Session 4 | 9
  Session 5 | 8
  Session 6 | 8

4. Primary Outcome: Rate of Delivery of Intervention Materials and Resources (Feasibility)
Description: 100% of intervention materials and resources are delivered as planned to intervention participants.
Time Frame: During the 12-week yoga intervention
Population: Compute the percentage of intervention participants who receive the materials and resources throughout the intervention. The number of participants analyzed was 33 because this outcome was measured during the 12-week yoga intervention and prior to the post-intervention data collection milestone. There were originally 34 participants randomized to the yoga intervention, but 1 intervention participant officially withdrew from the study prior to the start of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group
Number analyzed (Participants) | 33
Participants
  Yoga Equipment | 31
  Resource Guide | 33
  Pose Book | 33
  Facebook Group Invitation | 25
  Workshop Pamphlet | 28
  Workshop Book | 27

5. Primary Outcome: Rating of Assessment Measures (Feasibility)
Description: At least 80% intervention and control participants rate the assessments as not too burdensome (rated 1 or 2) on a scale from 1 (not burdensome) to 5 (very burdensome).
Time Frame: Baseline
Population: These survey items were sent via email to participants after baseline assessments were completed and prior to randomization. A total of 44 participants (25 intervention participants and 19 control group participants) completed the survey. Thus, the total sample size for this outcome measure is 44.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 25 | 19
Participants
  Traveling to the clinic to complete measurements | 20 | 15
  Getting weight and blood pressure measured by research staff | 21 | 17
  Completing electronic survey on an iPad | 23 | 16
  Collecting saliva samples for two days | 11 | 8
  Wearing the activity monitor for seven days | 19 | 14
  Traveling to the clinic to return saliva samples and activity monitor | 18 | 15

6. Primary Outcome: Completion of Assessment Measures (Feasibility)
Description: At least 90% intervention and control participants will complete baseline assessments.
Time Frame: Baseline
Population: Total sample of participants who enrolled, consented, and were randomized into the intervention and control groups. Excludes participant who withdrew from the study prior to randomization (n = 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 34 | 34
Participants
  Survey | 34 | 34
  Height, Weight, and Blood Pressure | 34 | 34
  ActivPAL Activity Monitor | 32 | 32
  Saliva Samples | 32 | 32

7. Primary Outcome: Rating of Assessment Measures (Feasibility)
Description: as for outcome 5
Time Frame: Post-intervention (within 2 months)
Population: At post-intervention, 57 participants completed a survey during in-person data collection that included 3 items rating burden of 1) traveling to the clinic, 2) getting weight and blood pressure measured, and 3) completing survey. The remaining 3 items rating burden of 1) collecting saliva samples, 2) wearing activity monitor, and 3) returning equipment were sent via email to participants after they returned their equipment. Only 6 participants responded to the 3 survey items from the email.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 31 | 26
Participants
  Traveling to the clinic to complete measurements | 27 | 19
  Getting weight and blood pressure measured by research staff | 30 | 22
  Completing electronic survey on an iPad | 25 | 20
  Collecting saliva samples for two days: number analyzed (Participants) | 4 | 2
  Collecting saliva samples for two days | 2 | 0
  Wearing the activity monitor for seven days: number analyzed (Participants) | 4 | 2
  Wearing the activity monitor for seven days | 3 | 1
  Traveling to the clinic to return saliva samples and activity monitor: number analyzed (Participants) | 4 | 2
  Traveling to the clinic to return saliva samples and activity monitor | 3 | 1

8. Primary Outcome: Completion of Assessment Measures (Feasibility)
Description: At least 90% of intervention and control participants will complete post-intervention assessments.
Time Frame: Post-Intervention (within 2 months)
Population: Excludes 1 intervention group participant who withdrew from the study after randomization but prior to start of the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 33 | 34
Participants
  Survey | 31 | 26
  Weight and Blood Pressure | 31 | 26
  ActivPAL Activity Monitor | 27 | 23
  Saliva Samples | 27 | 24

9. Primary Outcome: Rating of Assessment Measures (Feasibility)
Description: as for outcome 5
Time Frame: 3-month follow-up
Population: The total sample of participants (n = 51) who completed the survey during their 3-month follow-up data collection visit. The sample size for 2 of the survey items is n = 50 due to missing responses (i.e., the participant completed the rest of the survey but did not submit a response to that item).
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 23 | 28
Participants
  Traveling to the clinic to complete measurements | 17 | 17
  Getting weight and blood pressure measured by research staff | 20 | 27
  Completing electronic survey on an iPad | 17 | 21
  Collecting saliva samples for two days: number analyzed (Participants) | 22 | 28
  Collecting saliva samples for two days | 15 | 13
  Wearing the activity monitor for seven days | 14 | 22
  Traveling to the clinic to return saliva samples and activity monitor: number analyzed (Participants) | 23 | 27
  Traveling to the clinic to return saliva samples and activity monitor | 16 | 15

10. Primary Outcome: Completion of Assessment Measures (Feasibility)
Description: At least 90% of intervention and control participants will complete 3-month follow-up assessments.
Time Frame: 3-month follow-up
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 33 | 34
Participants
  Survey | 23 | 28
  Weight and Blood Pressure | 23 | 28
  ActivPAL Activity Monitor | 22 | 28
  Saliva Samples | 20 | 27

11. Primary Outcome: Rating of Intervention Components (Acceptability)
Description: At least 90% intervention participants rate the various intervention components (e.g., location, in-person classes, instructors, home-based resources) as acceptable with a rating of 4, 5, or 6 on a scale from 1 (strongly dislike) to 6 (strongly like).
Time Frame: Post-intervention (within 2 months)
Population: Of the 33 participants who were randomized to the yoga intervention group, 2 participants were lost to follow-up and did not complete the post-intervention survey that included items rating the acceptability of the intervention components. Thus, the sample size for this outcome measure is n = 31.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group
Number analyzed (Participants) | 31
Participants
  Intervention location: number analyzed (Participants) | 30
  Intervention location | 26
  Instructors | 31
  Yoga poses and sequencing (i.e., level of difficulty and modifications) | 29
  Yoga instruction (including music and use of Sanskrit/English terms) | 30
  Yoga equipment (i.e., mats, blocks, bolster, strap, blanket) | 31
  Availability of different class formats (i.e., in person, Zoom, recordings) | 29
  Class frequency of 3 times per week | 30
  Class time of day | 23
  Duration of the class (60 minutes) | 29
  Sharing circle at the end of each yoga class | 27
  Time of year of intervention (during the summer) | 23
  Biweekly workshops | 27
  Workshop resources (book and pamphlet) | 31
  Pose book | 31
  Private Facebook group and posts | 25

12. Primary Outcome: Participant Rating of Yoga Intervention (Acceptability)
Description: At least 90% intervention participants rate intervention acceptable (i.e., rating of 4, 5, or 6 on a scale from 1 (strongly dislike) to 6 (strongly like)) and enjoyable (i.e., rating of 3, 4, or 5 on a scale from 1 (not enjoyed) to 5 (enjoyed very much)).
Time Frame: Post-intervention (within 2 months)
Population: Of the 33 participants who were randomized to the yoga intervention group, 2 participants were lost to follow-up and did not complete the post-intervention survey that included items rating the acceptability of the intervention. Thus, the sample size for this outcome measure is n = 31.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group
Number analyzed (Participants) | 31
Participants
  Overall acceptability of yoga program | 30
  Enjoyment of program | 31

13. Primary Outcome: Number of Adverse Events (Safety)
Description: Zero adverse events (causes major disruption to participants' life, e.g., sprain, broken bone, cardiovascular event, death), zero moderate adverse events (causes minor inconvenience to participant, e.g., fainting spell, sore muscles for more than 3 days) and less than 10% of participants report mild adverse events (no major impact, e.g., headache, sore muscles for 2-3 days)
Time Frame: During the 12-week yoga intervention
Population: Of the 33 participants who were randomized to the yoga intervention group, 2 participants were lost to follow-up and did not attend any of the yoga sessions. Thus, the sample size for this outcome measure is n = 31. We did not assess Adverse Events within the control group during the course of the 12-week yoga intervention, as we did not have contact with the control group during this time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | Yoga Intervention Group
Number analyzed (Participants) | 31
Participants
  Adverse event (causes major disruption to participants' life) | 0
  Moderate adverse events (causes minor inconvenience to participant) | 0
  Mild adverse events (no major impact) | 1

14. Secondary Outcome: Sedentary Behavior
Description: Objective sedentary time (i.e., time spent sitting and lying down) assessed with activPAL4 micro accelerometer. Analyze data to report average total hours of sedentary behavior per day.
Time Frame: Seven consecutive days at three time points: baseline before intervention, post-intervention (within 2 months), and 3-month follow-up.
Population: At each time point, results will be reported for participants who returned activPAL4 micro accelerometers with monitor wear data. At baseline, 32 yoga intervention group participants and 32 control group participants returned activPAL4 micro accelerometers with monitor wear data.
Measure: Mean (Standard Deviation); unit: hours of sedentary behavior per day
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 32 | 32
hours of sedentary behavior per day
  Baseline | 10.7 (1.7) | 10.2 (2.0)
  Post-Intervention: number analyzed (Participants) | 27 | 23
  Post-Intervention | 11.4 (1.9) | 10.3 (1.8)
  3-Month Follow-Up: number analyzed (Participants) | 22 | 27
  3-Month Follow-Up | 10.8 (1.8) | 10.2 (2.4)

15. Secondary Outcome: Systolic and Diastolic Blood Pressure
Description: Measured using the automated OMRON Hem 907XL blood pressure recorder. Three blood pressures will be collected and averaged at each data collection time point following a two minute period of rest.
Time Frame: Three blood pressures will be collected and averaged at each of the 3 data collection time points (baseline, post-intervention (within 2 months), and 3 month follow-up)
Population: Blood pressure measures are missing from participants who did not complete in-person data collection visits at the post-intervention and 3-month follow-up time points, and from one intervention group participant who was unable to provide accurate blood pressure readings at both baseline and 3-month follow-up due to equipment malfunction.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 34 | 34
mmHg
  Baseline: Systolic Blood Pressure: number analyzed (Participants) | 33 | 34
  Baseline: Systolic Blood Pressure | 114.2 (13.6) | 116.1 (14.0)
  Baseline: Diastolic Blood Pressure: number analyzed (Participants) | 33 | 34
  Baseline: Diastolic Blood Pressure | 77.2 (11.5) | 77.2 (12.7)
  Post-Intervention: Systolic Blood Pressure: number analyzed (Participants) | 31 | 26
  Post-Intervention: Systolic Blood Pressure | 118.0 (18.4) | 115.9 (15.5)
  Post-Intervention: Diastolic Blood Pressure: number analyzed (Participants) | 31 | 26
  Post-Intervention: Diastolic Blood Pressure | 77.2 (11.7) | 75.6 (12.3)
  3-Month Follow-Up: Systolic Blood Pressure: number analyzed (Participants) | 22 | 28
  3-Month Follow-Up: Systolic Blood Pressure | 118.6 (16.1) | 119.6 (18.4)
  3-Month Follow-Up: Diastolic Blood Pressure: number analyzed (Participants) | 22 | 28
  3-Month Follow-Up: Diastolic Blood Pressure | 78.0 (12.4) | 78.0 (15.5)

16. Secondary Outcome: Perceived Stress
Description: Measured using the 14-item Perceived Stress Scale. Each item is scored from 1-5, with higher scores indicating higher perceived stress. Estimates represent the mean total score of the 14 items, ranging from 1-5. Scale was included in an online survey that participants completed at the data collection site via an iPad. Survey items asked participants how often they had experienced acute stress within last month.
Time Frame: Surveys will be distributed at each data collection timepoint (baseline, post-intervention (within 2 months), and 3 month follow-up)
Population: All participants who completed Perceived Stress Scale as part of the survey that was distributed at the in-person data collection time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Yoga Intervention Group | Control Group
Number analyzed (Participants) | 34 | 34
score on a scale
  Baseline | 2.9 (0.4) | 2.8 (0.5)
  Post-Intervention: number analyzed (Participants) | 31 | 26
  Post-Intervention | 2.6 (0.4) | 2.6 (0.5)
  Follow-Up: number analyzed (Participants) | 23 | 28
  Follow-Up | 2.7 (0.5) | 2.7 (0.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Intervention group participants were instructed to call their healthcare provider and notify the research staff if they experienced an injury or any adverse event. Participants in the Control Group were not assessed for deaths or adverse events.
Arm/Group | Yoga Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga Intervention Group (N=33)
Mild Adverse Event (Musculoskeletal and connective tissue disorders) | 1 (1) — Knee pain experienced during a yoga session.

LIMITATIONS AND CAVEATS:
Although Specific Aim 4 addressing the feasibility of salivary sample collection was achieved, due to budgetary constraints, the research team was unable to analyze the cortisol levels of the saliva samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT04710979/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04710979/ICF_001.pdf